CLINICAL TRIAL: NCT03065426
Title: Mechanisms That Predict Weight Trajectory After Bariatric Surgery: The Interactive Roles of Behavior and Biology
Brief Title: Microbiome and Bariatric Surgery
Acronym: Biobehavioral
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: North Dakota State University (Other)
Collaborators: Neuropsychiatric Research Institute (Unknown); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kristine Steffen, Associate Professor, North Dakota State University
Other Study IDs: BIO-XXX
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Weight Change, Body
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Roux-en-Y Gastric Bypass: Patients planning to undergo Roux-en-Y Gastric Bypass will be invited to participate in this study.
- Sleeve Gastrectomy: Patients planning to undergo Sleeve Gastrectomy will be invited to participate in this study.

SUMMARY:
This is a prospective, 24-month, longitudinal study of patients planning to undergo bariatric surgery (Roux-en-Y Gastric Bypass or Sleeve Gastrectomy) in which we aim to identify correlates and predictors of observed weight loss trajectories following bariatric surgery. This approach will expand current knowledge by examining the combined impact of empirically supported behavioral and biological data in a large sample over time. Intensive measurement of problematic eating behaviors, mood, and compliance with diet and exercise regimens post-surgery will be analyzed in the context of lterations in parallel with, or in response to, changes observed in the gut microbiota. Identifying these post-surgical predictors of weight loss and comorbidity resolution will allow for the development of individualized interventions to optimize surgery-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. In evaluation for Roux-en-Y Gastric Bypass or Sleeve Gastrectomy.
2. Age 18-65, inclusive

Exclusion Criteria:

1. Alcohol or substance use disorder in past year
2. Severe psychiatric disorder that may affect ability to complete the protocol
3. Regular tobacco use during the last year
4. Current medication taken routinely and known to impact factors that may affect the gut microbiome
5. Use of any oral or injectable antibiotic in the past month
6. Use of commercially available pre/pro biotic in the past month
7. History of significant disease/disorder that would be expected to impact the microbiome of the gut
8. Inability to engage in physical activity or dietary monitoring
9. Nonprescribed/illicit drug use
10. Pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants planning to undergo Roux-en-Y Gastric Bypass or Sleeve Gastrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2017-05-11 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Weight trajectory | 24 months
  Weight outcomes following bariatric surgery

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Neuropsychiatric Research Institute, Fargo, North Dakota
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
To the extent required by NIH and permitted by appropriate laws and rules. It will be available after the conclusion of the study and when the data have been cleaned.

REFERENCES:
- [Derived] Carroll I, Qian Y, Sorgen A, Steffen K, Heinberg L, Reed K, Malazarte A, Fodor A. Intestinal energy harvest is associated with post-bariatric surgery weight loss. Res Sq [Preprint]. 2024 Mar 29:rs.3.rs-4031151. doi: 10.21203/rs.3.rs-4031151/v1. PMID 38586018